CLINICAL TRIAL: NCT05194072
Title: A Phase 1 Study of Felmetatug Vedotin/SGN-B7H4V in Advanced Solid Tumors
Brief Title: A Study of Felmetatug Vedotin/SGN-B7H4V in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated for strategic reasons. The decision was not based on any safety and/or efficacy concerns
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNB7H4V-001; C5761001 (Other: Alias Study Number); 2023-503389-22-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms; Triple Negative Breast Neoplasms; HER2 Negative Breast Neoplasms; Hormone Receptor Positive Breast Neoplasms; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung; Cholangiocarcinoma; Gallbladder Carcinoma; Adenoid Cystic Carcinoma
Keywords: High-grade serous epithelial ovarian cancer; Primary peritoneal cancer; Fallopian tube cancer; HER2-negative breast cancer; HR positive breast cancer; Triple-negative breast cancer; TNBC; Endometrial carcinoma; Non-small cell lung cancer; NSCLC; SqCC; AC; ACC; Pfizer; Seattle Genetics
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms; Triple Negative Breast Neoplasms; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung; Cholangiocarcinoma; Gallbladder Neoplasms; Carcinoma, Adenoid Cystic | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Felmetatug Vedotin (Parts A, B, and C) (Experimental): Felmetatug Vedotin monotherapy
  Interventions: Drug: Felmetatug Vedotin
- Felmetatug Vedotin and Pembrolizumab (Parts D and E) (Experimental): Felmetatug Vedotin in combination with Pembrolizumab.
  Interventions: Drug: Felmetatug Vedotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Felmetatug Vedotin — Given into the vein (IV; intravenously)
  Other Names: SGN-B7H4V; PF-08046048
Drug: Pembrolizumab — 400 mg every 6 weeks, given by IV
  Other Names: Keytruda
  Arms: Felmetatug Vedotin and Pembrolizumab (Parts D and E)

SUMMARY:
The purpose of the study is to test the safety of the medicine called Felmetatug Vedotin alone and with pembrolizumab in participants with solid tumors. It will also look at the side effects of this medicine. A side effect is anything a medicine does to the body besides treating the disease.

This study is seeking for participants who either have cancer:

* that has spread in the body near where it started (locally advanced) and cannot be removed (unresectable),
* has spread through the body (metastatic), or have some cancer left over after surgery.

This study will have five parts.

* Parts A and B of the study will find out how much Felmetatug Vedotin should be given to participants.
* Part C will use the amount found in Parts A and B to find out how safe Felmetatug Vedotin is and if it works to treat solid tumor cancers.
* Part D will find out if and how much Felmetatug Vedotin can be given with pembrolizumab.
* Part E will use the amount found in Part D to find out how safe Felmetatug Vedotin with pembrolizumab is and if it works to treat triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

For Parts A, B, and C:

* Participants must have one of the following histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumor types:

  * High-grade serous epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer
  * HER2-negative, HR positive breast cancer
  * Triple-negative breast cancer (TNBC)
  * Endometrial carcinoma
  * Non-small cell lung cancer (Squamous cell carcinoma [SqCC], Adenocarcinoma [AC])
  * Cholangiocarcinoma or gallbladder carcinoma
  * Adenoid cystic carcinoma (ACC) For Part D: Participants must have histologically or cytologically confirmed locally advanced unresectable or metastatic TNBC.

For Part E:

* Cohort E1: Participants must have histologically or cytologically confirmed locally advanced unresectable or metastatic TNBC and must have CPS≥10 by local testing
* Cohort E2: Participants must have histologically or cytologically confirmed locally advanced unresectable or metastatic TNBC and must have CPS<10 by local testing
* Cohort E3: Participants must have triple negative breast cancer with residual disease following neoadjuvant therapy and definitive surgery

  * Parts A and B: Participants must have disease that is relapsed or refractory or be intolerant to SOC therapies, and, in the judgement of the investigator, should have no appropriate SOC therapeutic option
  * Part C: Participants must have disease that is relapsed or refractory or be intolerant to SOC therapies.
  * Part D and E1/E2: Participants must have had no prior treatment for locally advanced unresectable or metastatic TNBC
  * Part E3: Participants must have completed at least 6 cycles of neoadjuvant therapy for locally advanced unresectable or metastatic TNBC
  * Tumor tissue is required for enrollment.
  * Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
  * Measurable disease per RECIST version 1.1 at baseline (not applicable for E3 participants).

Exclusion Criteria:

* History of another malignancy within 3 years before the first dose of study drug. Any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death.
* Known active central nervous system metastases. Participants with previously treated brain metastases may participate provided they:

  * are clinically stable for at least 4 weeks prior to study entry after brain metastasis treatment
  * have no new or enlarging brain metastases
  * and are off corticosteroids prescribed for symptoms associated with brain metastases for at least 7 days prior to the first dose of study treatment.
* Carcinomatous meningitis
* Previous receipt of an MMAE-containing agent or an agent targeting B7-H4
* Pre-existing neuropathy ≥ Grade 2 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
* Corneal disease or injury requiring treatment or active monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30 days after last study treatment, up to approximately 5 years
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Number of participants with laboratory abnormalities | Through 30-37 days after last study treatment, up to approximately 5 years
Number of participants with dose limiting toxicities (DLTs) | Up to 28 days
Number of participants with dose limiting toxicities (DLTs) and overall safety by dose level | Through 30-37 days after last study treatment; up to approximately 5 years

SECONDARY OUTCOMES:
Confirmed objective response rate (ORR) by investigator assessment | Up to approximately 5 years
  The proportion of participants with complete response (CR) or partial response (PR) which is subsequently confirmed as assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 by investigator.
Complete response rate (CRR) | Up to approximately 5 years
  The proportion of participants achieving a CR as determined by the investigator per RECIST Version 1.1.
Duration of response (DOR) | Up to approximately 5 years
  The time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression or to death due to any cause.
Progression-free survival (PFS) | Up to approximately 5 years
  The time from the start of any study treatment to first documentation of disease progression or to death due to any cause.
Invasive disease-free survival (iDFS) | Up to approximately 5 years
  The time from the start of any study treatment until the date of first occurrence of one of the following events: ipsilateral invasive breast tumor (local) recurrence, regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and skin of ipsilateral breast), or distant (metastatic) recurrence; contralateral invasive breast cancer; second primary non-breast invasive cancer (other than squamous of basal cell skin cancer); or death from any cause.
Pharmacokinetic (PK) parameter - Area under the curve (AUC) | Through 30-37 days after last study treatment; up to approximately 3 years
  To be summarized using descriptive statistics.
PK parameter - Maximum concentration (Cmax) | Through 30-37 days after last study treatment, up to approximately 3 years
  To be summarized using descriptive statistics.
PK parameter - Time to maximum concentration (Tmax) | Through 30-37 days after last study treatment, up to approximately 3 years
  To be summarized using descriptive statistics.
PK parameter - Apparent terminal half-life (t1/2) | Through 30-37 days after last study treatment, up to approximately 3 years
  To be summarized using descriptive statistics.
PK parameter - Trough concentration (Ctrough) | Through 30-37 days after last study treatment, up to approximately 3 years
  To be summarized using descriptive statistics.
Incidence of antidrug antibodies (ADAs) | Through 30-37 days after last study treatment, up to approximately 3 years
  To be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (20):
  - UCHealth Sue Anschutz-Rodgers Eye Center, Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - Presbyterian/St Lukes Medical Center, Denver, Colorado
  - AdventHealth Celebration Infusion Center, Celebration, Florida
  - AdventHealth Medical Group Oncology Research at Celebration, Celebration, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Community Health Network, Inc., Indianapolis, Indiana
  - START Midwest, Grand Rapids, Michigan
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center Investigational Pharmacy Services, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada
- Hamato-Onkologische Phase 1 Unit der Charite/Charite Research Organisation, Berlin, Germany
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - START Madrid-Hospital Universitario HM Sanchinarro, Madrid
- Sarah Cannon Research Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNB7H4V-001